CLINICAL TRIAL: NCT01065493
Title: QuitAdvisorMD: A Point-of-care Tool for Brief Smoking Cessation Interventions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Silverchair Science & Communications, LLC (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44DA026682 (NIH); R44DA026682 (NIH)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Smoking; Tobacco Use Disorder
MeSH Terms: conditions — Smoking; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Software Assisted Lifestyle Counseling (Experimental)
  Interventions: Other: QuitAdvisorMD Software Algorithm
- Lifestyle Counseling (Active Comparator): Status quo smoking cessation counseling.
  Interventions: Behavioral: Standard Smoking Cessation Counseling

INTERVENTIONS:
Other: QuitAdvisorMD Software Algorithm — QuitAdvisorMD, a set of brief clinical assessments, counseling scripts and intervention instruments for smoking cessation in primary care settings
  Arms: Software Assisted Lifestyle Counseling
Behavioral: Standard Smoking Cessation Counseling — Standard Smoking Cessation Counseling
  Arms: Lifestyle Counseling

SUMMARY:
QuitAdvisorMD: A point-of-care tool for brief smoking cessation interventions Under a Phase II SBIR grant supported by NIH/NIDA, we are developing QUITAdvisorMD: a point-of-care, patient-centered resource for counseling patients who smoke or use tobacco products. It is based on the principles of Motivational Interviewing, a non-confrontational and very effective method for intervening and treating these patients; the 5 A's of behavioral interventions; and the Transtheoretical Model of Change. Through a point and click interface, the tool uses a series of interview questions designed to motivate patients to stop smoking by first assessing their stage of change and then offering effective stage-based interventions and interview techniques. The tool also offers stage-tailored patient information, a clinician educational reference, and the ability to communicate support information patients via email and/or text message.

ELIGIBILITY:
Inclusion Criteria:

* any physician providing care for members of Southern Health through primary care and have access to a point-of-care computing device (Smartphone, desktop PC, etc) during patient visits.

Exclusion Criteria:

* Lack of appropriate computing device

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
The goal of the evaluation is to assess the ability of QuitAdvisorMD to influence smoking cessation as measured by the primary outcome of the increase in physician initiated smoking cessation counseling. | 12 Months

SECONDARY OUTCOMES:
Secondary outcomes will include, 1) the increase in ability of clinicians to provide appropriate stage-based smoking cessation assistance, and 2) the increase in patient quit attempts. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: George Reynolds, BA, Principal Investigator — Silverchair, Inc; Scott Strayer, MD, Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States